CLINICAL TRIAL: NCT06071013
Title: A Phase I/Phase II Study of Nintedanib Plus EGFR TKI In EGFR-mutated Non-small Cell Lung Cancer Patients
Brief Title: Nintedanib Plus EGFR TKI In EGFR-mutated Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH112-REC2-121
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Non-small Cell Lung Cancer; EGFR Gene Mutation; EGFR-TKI Resistant Mutation
Keywords: nPKC delta; Angiogenesis; EGFR TKI drug resistant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib; Gefitinib; Erlotinib Hydrochloride; Afatinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nintedanib + gefitinib/erlotinib/afatinib/osimertinib (Experimental): Nintedanib will administered orally twice per day Gefitinib will administered orally once daily Erlotinib will administered orally once daily Afatinib will administered orally once daily Osimertinib will administered orally once daily
  Interventions: Drug: Nintedanib, gefitinib, erlotinib, afatinib, osimertinib

INTERVENTIONS:
Drug: Nintedanib, gefitinib, erlotinib, afatinib, osimertinib — Nintedanib is a multiple tyrosine kinase inhibitor that can bind competitively to the ATP-binding pocket of these receptors and block intracellular signaling, which is critical for the proliferation and migration.
  Gefitinib, erlotinib and afatinib are the first- and second- generation of EGFR tyrosine kinase inhibitors that reversibly and irreversibly inhibit the binding of ATP to the phosphate-binding loop of ATP binding site in the kinase domain of EGFR, leading to the inhibition of cell proliferation and induction of apoptosis of cancer cells.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nintedanib with EGFR-TKI in participants with advanced EGFR-TKI-resistant non-small cell lung cancer

DETAILED DESCRIPTION:
The efficacy of the regimen is evaluated by participants' progression-free survival and overall survival.

Nintedanib is a medication that blocks endothelial cells in tumor microenvironments and is effective in delaying tumor progression. Nintedanib is also a drug approved for idiopathic pulmonary fibrosis in the clinic.

The participants will take 1 nintedanib tablet after a meal twice per day with a twelve-hour interval. EGFR TKI-gefitinib, erlotinib, afatinib, or osimertinib will be taken 1 tablet once per day during each treatment cycle. The treatment cycle in this study is 30 days.

In this study, the participants will have a physical exam in 6 weeks and 12 weeks after the initiation of the treatment. In the 6 weeks of the study, the participants will have blood tests and a CT scan. About 5cc of blood will be collected each time. In addition, the participant's tumor will be measured by a CT scan every 12 weeks.

If the participants develop any unacceptable symptoms or changes in liver function tests, the participants' treatment may be delayed and/or the dose decreased until the symptoms are disappeared. It may even be necessary to stop your treatment. The doctor will inform the participant of any changes in the participants' treatment schedule or in the doses of medication after he/she evaluates the participants in the clinic.

After treatment ends, the participants will have a follow-up visit at the clinic. At this visit, the participants will have a complete physical exam, including blood (about 5cc) tests and CT scan to measure the size of the tumors.

This is an investigational study. Up to 20 participants will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 20 to 70 years old, are pathologically confirmed advanced (stage III and IV) non-small cell lung cancer.
2. Positive EGFR mutations are diagenesis.
3. Participants with histologically/cytologically confirmed locally advanced or metastatic adenocarcinoma subtype NSCLC after the failure of first-line EGFR tyrosine kinase inhibitors- gefitinib, erlotinib, afatinib, or osimertinib.
4. Participants must have adequate hepatic, renal, and bone marrow function

Exclusion Criteria:

1. Participants previously received first-line EGFR tyrosine kinase inhibitor with serious side effects.
2. Participants have known hypertension, and chronic liver and gastrointestinal disease.
3. Participants have known brain metastasis.
4. Female participants who are pregnant or breast-feeding
5. Participants have a known diagnosis of negative nPKCδ expression by immunohistochemistry (IHC).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
The toxicity of combinate nintedanib and EGFR TKI | Assessed every 6 weeks of chest CT scan until PD.
Patient objective response rate | Assessed every 6 weeks of chest CT scan

SECONDARY OUTCOMES:
Overall survival | Assessed every 12 weeks thereafter up to end of study at approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pulmonary Medicine, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan